CLINICAL TRIAL: NCT04579627
Title: How Has the Increased Use of FFP3 Style Respirators During the COVID-19 Pandemic Affected Hospital Doctor's Facial Hair? Implications for Staff Safety and Welfare.
Brief Title: Facial Hair, PPE and COVID-19
Acronym: FACIAL HAIR
Status: Completed | Type: Observational
Sponsor: Royal Cornwall Hospitals Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 283609
Record Dates: First submitted 2020-10-06; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-06

CONDITIONS: COVID; Safety Issues
Keywords: Facial Hair; Beard; Personal Protective Equipment
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospital Doctors: Hospital doctors working at Royal Cornwall Hospital during the COVID-19 pandemic
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — A single survey questionnaire to staff to report their demographics and facial hair styles between January and April 2020

SUMMARY:
An observational cross sectional questionnaire study looking into facial hair of hospital doctors during the COVID-19 pandemic, and how personal protective equipment guidance has affected this.

DETAILED DESCRIPTION:
COVID-19 is a highly contagious virus which has caused a global pandemic. There have been significant health consequences for healthcare workers, which may be related to the provision of personal protective equipment (PPE). Following PPE guidance is a significant health and safety concern, under which facial hair guidance for tight fitting masks falls.

This has implications as FFP3 masks are not the only form of PPE for the face, and this study may highlight a need for employers to diversify which PPE they supply to their employees, such as full hoods if staff need to maintain facial hair for cultural or religious reasons.

As such, facial hair has potential implications for patient safety, but also these have to be balanced with personal or religious reasons for maintaining facial hair. Our study aimed to determine the facial hair styles of hospital doctors, and reasons for maintaining them during the COVID-19 pandemic. We also looked at whether these styles adhered to the PPE guidance set about by Public Health England (PHE)

ELIGIBILITY:
Inclusion Criteria:

All hospital doctors working at the main site at Royal Cornwall Hospital between January and April 2020 were included in the study population. This includes all genders and ethnicities.

Exclusion Criteria:

The principle exclusion criteria were those who did not work at the Royal Cornwall Hospital main site. Also, while not forming part of the exclusion criteria, those who are unable to grow facial hair were excluded from the statistical analyses.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All hospital doctors working at Royal Cornwall Hospital between January 2020 and April 2020.
Sampling Method: Non-Probability Sample
Enrollment: 358 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-06-08 (Actual)

PRIMARY OUTCOMES:
Change in facial hair between January 2020 and during April 2020. | January 2020 and during April 2020.
  Our primary outcome measure was change in facial hair between January 2020 (before guidance was circulated in the UK about facial hair), and during April 2020 (after guidance was circulated relating to PPE appropriate facial hair)

SECONDARY OUTCOMES:
Does facial hair change adhere to the PPE guidance from PHE | January 2020 and during April 2020.
  Does facial hair change adhere to the PPE guidance from PHE

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Cornwall Hospital, Truro, Cornwall, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Informed Consent Form (2020-05-05): https://cdn.clinicaltrials.gov/large-docs/27/NCT04579627/ICF_000.pdf
  • Study Protocol (2020-05-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT04579627/Prot_001.pdf